CLINICAL TRIAL: NCT03380858
Title: REINFORCEMENT ANASTOMOSIS IN ONCOLOGIC COLORECTAL SURGERY
Brief Title: REINFORCEMENT ANASTOMOSIS WITH Modified Cyanacrylate IN Patients Undergoing to Oncologic Colorectal Surgery With Colorectal Anastomosis
Acronym: ANASTOSEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Daniela Rega, doctor, National Cancer Institute, Naples
Other Study IDs: 04/17oss
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: colectomy — colectomy resection

SUMMARY:
In colorectal surgery about 30% of postoperative mortality is attributed to anastomotic leak, whit an incidence range between 1.8% and 15.9%. Preventing the anastomotic leak can therefore bring benefits to the patient and the health system. To date we have technologically advanced suturizers and the correct realization (well-vascularized margins, not in tension, etc.) remains crucial to prevent anastomotic dehiscence. Experimental results demonstrate that modified cyanacrylate is a suitable potential "reinforcement" on intestinal anastomoses (manual or linear intra-corporeal). Applied after mechanical anastomosis, it polymerizes in a short time, closing the spaces of the suture line between one point and the other, expressing an adhesive, hemostatic and sealing action on the tissues, also creating an effective antiseptic barrier towards of the most common infectious or pathogenic agents.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* patients undergoing to oncologic colorectal surgery with colorectal anastomosis

Exclusion Criteria:

* refuse informed consent
* patients undergoing to oncologic colorectal surgery without colorectal anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 390 consecutive patients undergoing colorectal resective surgery with intestinal anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2019-05-02 (Estimated)

PRIMARY OUTCOMES:
fistula incidence | From day of surgery up to 30 postoperative days

SECONDARY OUTCOMES:
anastomitic bleeding | From day of surgery up to 30 postoperative days
infection | From day of surgery up to 30 postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Pascale, Napoli, Italy